CLINICAL TRIAL: NCT03473470
Title: Evaluation of the Active Warming Effects on Maternal and Neonatal Outcomes During Cesarean Delivery
Brief Title: Evaluation of the Active Warming Effects on Maternal and Neonatal Outcome During Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, MD, University of Foggia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 76/CE/2017
Record Dates: First submitted 2018-02-27; First posted 2018-03-22 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Hypothermia; Anesthesia
Keywords: Maternal and Neonatal Hypothermia, cesarean delivery
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- not warmed (No Intervention): Not warming system
- warmed group 1 (Active Comparator): forced air warming and warmed intravenous fluids
  Interventions: Device: forced air warming and warmed intravenous fluids
- warmed group 2 (Active Comparator): warmed intravenous fluids
  Interventions: Device: warmed intravenous fluids

INTERVENTIONS:
Device: forced air warming and warmed intravenous fluids — Use of warming system (forced air)
  Arms: warmed group 1
Device: warmed intravenous fluids — Use of warming system to have warmed intravenous fluids
  Arms: warmed group 2

SUMMARY:
A prospective randomized study of healthy term parturients undergoing cesarean delivery was designed to assess the impact of the active warming on perioperative and postoperative temperature.

The main objective is to evaluate the maternal core temperature in the perioperative and postoperative period during cesarean delivery.

The secondary objectives are to assess the incidence of maternal hypothermia, the incidence of maternal shivers, the evaluation of maternal thermal comfort, the neonatal temperature at birth, the Apgar score at 1 and 5 minutes, the umbilical pH, the evaluation of coagulative assessment in case of maternal hypothermia trough the use of thromboelastography.

The patients are randomized into three groups: a group of no warmed patients, a second group of Active waming patients with iv fluids and lower body forced air warming and a third group of Active warming patients with only warmed iv fluids.

The inclusion criteria are healthy parturients up to age 18. The exclusion criteria included parturients who develop fever, diabetes mellitus, BMI up to 40kg/ m2, coagulative disorders, pre eclampsia or eclampsia, all the factors that can cause intraoperative bleeding such as placental abruption or antecedent placenta overgrowth ( placenta previa).

DETAILED DESCRIPTION:
The doctor's main purposes during the perioperative period are the monitorign and maintenance of normothermia, as well as the haemodynamic, respiratory, metabolic, analgesic control and monitoring.

Mild hypothermia ( core temperature between 36° and 33° C) is common during general, locoregional or blended anaesthesia. A mild hypothermia can cause a cardiovascular, haematological, metaolic and hormonal alterations that can explain an increased mortality and morbidity in hypothermia patients versus normothermia patients.

Thermic decrease is a physiological event during general or locoregional anaesthesia. Particularly spinal and epidural anaesthesia can cause the thermic decrease because of vasodilation below the level of the sensitive and neuroaxial blockade. In this way there is in the patient an increased heat loss trough radiation. The neuroaxial techniques can reduce the sensory connections and the level of vasoconstriction above the level of the sensorial blockade, reducing the patient capacity to maintain the poichilothermia.

The consequences of hypothermia are important because they can influence the intraoperative management causing complications extending the recovering time and the hospitalization.

The environmental temperature is a critical factor for the development of hypothermia , especially in critically patients. In order to avoid the deveopment of hypothermia the environmental temperature must be maintainde between 21° and 24° C and humidity level of 40- 60%.

Maternal hypothermia is common during cesarean delivery and it can exercise influence over neonatal temperature.

When a mother develops hypothermia the newborn can shows hypotheria, umbilical acidosis, low Apgar score at birth.

The recorded data are the demographic data of the patient such as weight, age and height, the vital signs such as heart rate, arterial pressure, SpO2 or EtCO2 during general anaesthesia, BMI, gestational age and parity, type of anaesthesia, doses and type of anaesthetic used, the development of adverse effects such as hypothermia or hypothension, the blood leaks, the environmental temperature on operative theatre, the temperature of fluids iv in the perioperative period, the maternal core temperature at preoperative, during induction of anaesthesia, after 5 minutes initiating anaesthesia, and then every 10 minutes until the end of the cesarean delivery and also at child birth, at the exit of operative theatre. Maternal temperature measurment will be obtained by using a skin sensor Spot On on a temporal region, the neonatal axillary temperature at 1 and5 minutes from birth using a digital thermometer, Apgar score and umbilical cord blood pH, the pain evaluation using a VAS scale ( 0-10), the maternal shivering by the Bedside Shivering Assessment scale, the maternal comfort using a verbal numerical scale ( 0 = as worst immaginable cold 50= as thermoneutral and 100= as insufferably hot), the timing of pain at induction of anaesthesia and then every 10 minutes until the operative room exit.

ELIGIBILITY:
Inclusion Criteria: all healthy parturients over eighteen years undergoing cesarean delivery

Exclusion Criteria:

* Fever;
* Diabetes mellitus;
* BMI> 40Kg/m²;
* Coaugulation disorders;
* Pre-eclampsia and eclampsia;
* Increased risk of intraoperative hemorrhage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2016-12-22 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
incidence of hypothermia (body temperature < 36°C) | From the date of randomization until the end of surgery, up to four hours of surgery
  to assess the incidence of maternal hypothermia during caesarean delivery

SECONDARY OUTCOMES:
Incidence of maternal shivering | From the date of randomization until the end of surgery, up to four hours of surgery
  Use of the Bedside shivering scale (score 0 no shiver, score 1 mild shiver at the neck or thorax, score 2 moderate shiver at the neck, thorax and arms, score 3 severe shiver at the neck, thorax, arms and legs. Score 2 and 3 are the worse outcomes
Neonatal body temperature (T°C) | From neonatal birth until five minutes after the birth
  with axillary thermometer
Neonatal Apgar score | From neonatal birth and until five minutes after the birth
  Measurement of Apgar score
Incidence of maternal coagulative disorders | From the date of randomization until the end of surgery, up to four hours of surgery
  Thromboelastography
maternal thermal comfort | From the date of randomization until the end of surgery, up to four hours of surgery
  Use of a VAS 0-100 scale (100=insufferably hot, 50=thermoneutral and 0=unimaginably cold); 50 thermoneutral is the better outcome cold, 0=thermally neutral, +50=insufferably hot

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Cotoia, MD, Principal Investigator — University of Foggia
Locations (1):
- Ospedali Riuniti, Foggia, Apulia, Italy

IPD SHARING:
Plan to Share IPD: No